CLINICAL TRIAL: NCT00811252
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Duloxetine-referenced, Fixed Dose Study Comparing the Efficacy and Safety of [Vortioxetine] Lu AA21004 in Acute Treatment of Major Depressive Disorder in Elderly Patients
Brief Title: Randomised Placebo-controlled Duloxetine-referenced Study of Efficacy and Safety of 5 mg of Vortioxetine (Lu AA21004) in Acute Treatment of Major Depressive Disorder in Elderly Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12541A; 2008-002901-38 (EudraCT Number)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Elderly; Acute treatment
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vortioxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vortioxetine 5 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Duloxetine 60 mg (Other): Active reference
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Placebo — capsules; daily; orally
  Arms: Placebo
Drug: Vortioxetine (Lu AA21004) — encapsulated tablets; daily; orally
  Other Names: Brintellix
  Arms: Vortioxetine 5 mg
Drug: Duloxetine — encapsulated tablets; daily; orally
  Other Names: Cymbalta®
  Arms: Duloxetine 60 mg

SUMMARY:
To assess the efficacy of Vortioxetine (5 mg daily) versus placebo in the acute treatment of depression by means of the change from baseline in the 24-item Hamilton Depression Scale (HAM-D24) total score after 8 weeks of double-blind treatment in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical Diagnosis of recurrent Major Depressive Episode (MDE) according the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria with:

* Reported duration of the current episode of at least 4 weeks
* MADRS total score >=26
* At least one previous MDE before the age of 60 years

Exclusion Criteria:

* Mini Mental State Exam (MMSE) <24
* Any current anxiety disorder as defined in the DSM-IV-TR
* Current or past history of manic or hypomanic episode, schizophrenia, or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR
* Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR
* Presence or history of a clinically significant neurological disorder (including epilepsy)
* Neurodegenerative disorder (Alzheimer's disease, Parkinson disease, multiple sclerosis, Huntington disease, etc)
* Any Axis II disorder that might compromise the study
* Significant risk of suicide according to the investigator's opinion, or has a score >=5 on item 10 of the MADRS or has made a suicide attempt in the previous 6 months

Other inclusion and exclusion criteria may apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 453 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Katona C, Hansen T, Olsen CK. A randomized, double-blind, placebo-controlled, duloxetine-referenced, fixed-dose study comparing the efficacy and safety of Lu AA21004 in elderly patients with major depressive disorder. Int Clin Psychopharmacol. 2012 Jul;27(4):215-23. doi: 10.1097/YIC.0b013e3283542457. PMID 22572889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were mainly recruited via psychiatric, psycho-geriatric, and geriatric inpatient or outpatient settings.
Pre-assignment Details: The study consisted of a Screening Period; an 8-week Core Treatment Period; a 1-week double-blind down-taper period (Week 9); and a 4-week Safety Follow-up Period after completion/withdrawal (Weeks 8 to 12).
Groups:
- Vortioxetine 5 mg; Duloxetine 60 mg: encapsulated tablets; daily; orally
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Started | 145 | 156 | 151
Completed | 128 | 136 | 128
Not Completed | 17 | 20 | 23
Not completed — Adverse Event | 6 | 10 | 15
Not completed — Lack of Efficacy | 7 | 2 | 0
Not completed — Protocol Violation | 3 | 3 | 2
Not completed — Withdrawal of Consent | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Administrative or Other Reasons | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Full-analysis set (FAS) - all patients in the all-patients-treated set (APTS) who had at least one valid post-baseline assessment of the primary efficacy variable
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 145 | 156 | 151 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (4.4) | 70.5 (4.8) | 70.9 (5.5) | 70.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 107 | 100 | 297
  Male | 55 | 49 | 51 | 155
HAM-D-24 [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
  units on a scale | 29.4 (5.1) | 29.2 (5.0) | 28.5 (4.9) | 29.0 (5.0)
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 30.3 (3.2) | 30.7 (3.6) | 30.4 (3.1) | 30.5 (3.3)
HAM-A [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
  units on a scale | 19.5 (5.7) | 19.9 (5.8) | 19.2 (6.5) | 19.5 (6.0)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 4.7 (0.7) | 4.8 (0.7) | 4.7 (0.8) | 4.7 (0.7)
GDS [Mean (Standard Deviation); unit: units on a scale] — The Geriatric Depression Scale (GDS) is a patient self-rating scale designed for the screening of depression in the elderly. It has also been validated as a measure of depression severity. The original version consists of 30 questions with a yes/no answer. In this study, the short 15-item version was used. The total score ranges from 0 to 15, with 15 representing maximum severity.
  units on a scale | 7.7 (2.0) | 7.4 (2.2) | 7.7 (2.3) | 7.6 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HAM-D-24 Total Score After 8 Weeks of Treatment
Description: The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: Full-analysis set (FAS) - all patients in the all-patients-treated set (APTS) who had at least one valid post-baseline assessment of the primary efficacy variable; last observation carried forward (LOCF); analysis of covariance (ANCOVA)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | -10.3 (0.76) | -13.7 (0.74) | -15.8 (0.75)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; As soon as an endpoint was non-significant at the 0.05 level of significance, the testing procedure was stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.0011, ANCOVA — Since p-value <0.05, hierarchically testing continued; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-5.31 to -1.34], Standard Error of Mean 1.01 — A statistical testing strategy was defined a priori for a single dose of vortioxetine that was tested versus placebo in the primary and key secondary efficacy analyses
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -5.48, 95% CI 2-sided [-7.50 to -3.46], Standard Error of Mean 1.03

2. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 6 Weeks of Treatment
Time Frame: Baseline and Week 6
Population: FAS; LOCF, ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | -10.2 (0.71) | -12.3 (0.69) | -14.4 (0.70)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0240, ANCOVA — Since p-value <0.05, hierarchically testing continued; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-3.98 to -0.28], Standard Error of Mean 0.94 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -4.22, 95% CI 2-sided [-6.10 to -2.34], Standard Error of Mean 0.96

3. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 4 Weeks of Treatment
Time Frame: Baseline and Week 4
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | -8.99 (0.64) | -10.1 (0.62) | -12.3 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.2134, ANCOVA — Since p-value >0.05, hierarchically testing stopped here; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-2.72 to 0.61], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -3.30, 95% CI 2-sided [-4.99 to -1.60], Standard Error of Mean 0.86

4. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 2 Weeks of Treatment
Time Frame: Baseline and Week 2
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | -6.66 (0.53) | -6.95 (0.51) | -7.91 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.6879, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.67 to 1.10], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0827, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-2.65 to 0.16], Standard Error of Mean 0.72

5. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 1 Week of Treatment
Time Frame: Baseline and Week 1
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 154 | 147
units on a scale | -3.62 (0.41) | -4.04 (0.40) | -3.48 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.4482, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.49 to 0.66], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.7971, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.95 to 1.24], Standard Error of Mean 0.56

6. Secondary Outcome: Change From Baseline in MADRS Total Score After 8 Weeks of Treatment
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | -11.2 (0.77) | -15.5 (0.75) | -18.0 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — A nominal p-value is provided. No correction for multiplicity was made; Mean Difference (Final Values) = -4.29, 95% CI 2-sided [-6.32 to -2.26], Standard Error of Mean 1.03

7. Secondary Outcome: Change From Baseline in HAM-A Total Score After 8 Weeks of Treatment
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | -5.74 (0.55) | -8.09 (0.54) | -9.28 (0.54)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.0015, ANCOVA — A nominal p-value is provided. No correction for multiplicity was made; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-3.80 to -0.91], Standard Error of Mean 0.74

8. Secondary Outcome: Change From Baseline in CGI-S Score After 8 Weeks of Treatment
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
Time Frame: Baseline and Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | -1.03 (0.11) | -1.63 (0.10) | -2.05 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — A nominal p-value is provided. No correction for multiplicity was made; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.88 to -0.32], Standard Error of Mean 0.14

9. Secondary Outcome: Change in Clinical Status Using CGI-I Score at Week 8
Description: The Clinical Global Impression - Global Improvement (CGI-I) is a 7-point scale rated from 1 (very much improved) to 7 (very much worse). The investigator rated the patient's overall improvement relative to baseline, whether or not, in the opinion of the investigator, this was entirely due to the drug treatment.
Time Frame: Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
units on a scale | 2.91 (0.10) | 2.35 (0.09) | 2.07 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — A nominal p-value is provided. No correction for multiplicity was made; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.82 to -0.31], Standard Error of Mean 0.13

10. Secondary Outcome: Change From Baseline in GDS Total Score After 8 Weeks of Treatment
Description: The Geriatric Depression Scale (GDS) is a patient self-rating scale designed for the screening of depression in the elderly. It has also been validated as a measure of depression severity. The original version consists of 30 questions with a yes/no answer. In this study, the short 15-item version was used. The total score ranges from 0 to 15, with 15 representing maximum severity.
Time Frame: Baseline and Week 8
Population: FAS; observed cases (OC); ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 144 | 154 | 142
units on a scale | -0.65 (0.17) | -1.08 (0.17) | -1.32 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.0552, ANCOVA — A nominal p-value is provided. No correction for multiplicity was made; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.88 to 0.01], Standard Error of Mean 0.23

11. Secondary Outcome: Proportion of Responders at Week 8 (Response Defined as a >=50% Reduction in the HAM-D-24 Total Score)
Time Frame: Week 8
Population: FAS; LOCF
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
percentage of patients | 35 | 53 | 63
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.0008, Regression, Logistic — A nominal p-value is provided. No correction for multiplicity was made; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.26 to 0.70]

12. Secondary Outcome: Proportion of Remitters at Week 8 (Remission Defined as a MADRS Total Score <=10)
Time Frame: Week 8
Population: FAS; LOCF
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 148
percentage of patients | 21 | 34 | 47
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.0090, Regression, Logistic — A nominal p-value is provided. No correction for multiplicity was made; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.27 to 0.83]

13. Secondary Outcome: Risk of Suicidality Using C-SSRS Scores
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) was developed by researchers at Columbia University as a tool to systematically assess suicidal ideation and behaviour in patients during participation in a clinical study. The C-SSRS is composed of questions that address suicidal behaviour and questions that address suicidal ideation, with sub-questions that assess severity. The tool was administered via an interview with the patient.
Time Frame: Up to 8 weeks
Population: C-SSRS Data by Columbia Classification Algorithm for Suicide Assessment (C-CASA) Category (APTS)
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Number analyzed (Participants) | 114 | 121 | 114
participants
  No ideation or behavior | 103 | 107 | 106
  Completed Suicide | 0 | 0 | 0
  Suicide Attempt | 0 | 0 | 1
  Preparatory Actions Toward Imminent Suicidal Behav | 0 | 0 | 0
  Suicidal Ideation: Passive | 8 | 14 | 7
  Suicidal Ideation: Active / Nonspecific | 3 | 0 | 0
  Suicidal Ideation: Active / Method, but no intent | 0 | 0 | 0
  Suicidal Ideation: Active / Method and intent, but | 0 | 0 | 0
  Suicidal Ideation: Active / Method, intent, and pl | 0 | 0 | 0
  Self-Injurious Behavior Without Suicidal Intent | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 8-week double-blind treatment period and 4-week safety follow-up period Other Adverse Events: 8-week double-blind treatment period
Arm/Group | Placebo | Vortioxetine 5 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 4/145 | 1/156 | 1/151
Other Adverse Events (participants affected / at risk) | 63/145 | 72/156 | 104/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=145) | Vortioxetine 5 mg (N=156) | Duloxetine 60 mg (N=151)
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/55 | 0/49 | 1/51
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=145) | Vortioxetine 5 mg (N=156) | Duloxetine 60 mg (N=151)
Constipation (Gastrointestinal disorders) | 6 | 10 | 21
Diarrhoea (Gastrointestinal disorders) | 10 | 8 | 14
Dry mouth (Gastrointestinal disorders) | 7 | 10 | 33
Nausea (Gastrointestinal disorders) | 12 | 34 | 50
Fatigue (General disorders) | 5 | 11 | 16
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 8
Dizziness (Nervous system disorders) | 10 | 14 | 14
Headache (Nervous system disorders) | 25 | 18 | 18
Somnolence (Nervous system disorders) | 3 | 4 | 16
Ejaculation delayed (Reproductive system and breast disorders) | 0/55 | 0/49 | 3/51
Erectile dysfunction (Reproductive system and breast disorders) | 0/55 | 0/49 | 3/51
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 6 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub-publications. H. Lundbeck A/S follows the Vancouver declaration with respect to authorship.